CLINICAL TRIAL: NCT02051413
Title: Beta-arrestins and Response to Venlafaxine in Major Depressive Disorder
Brief Title: Beta-arrestins and Response to Venlafaxine in Major Depressive Disorder (MDD) (DEPARRESTCLIN)
Acronym: DEPARRESTCLIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C13-25; 2013-004326-29 (EudraCT Number)
Record Dates: First submitted 2014-01-22; First posted 2014-01-31 (Estimated); Last update posted 2025-09-02 (Actual); Status verified 2021-08

CONDITIONS: Major Depressive Disorder; Major Depressive Episode
Keywords: Major depression; Antidepressant drug; Beta-arrestin; Biomarker; Predictive factor
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Venlafaxine extended release (Other): Venlafaxine extended-release, flexible dose
  Interventions: Drug: Venlafaxine extended release

INTERVENTIONS:
Drug: Venlafaxine extended release — antidepressant drug
  Other Names: EFFEXOR

SUMMARY:
Predictive factors and biomarkers of response to antidepressants in major depressive disorder are scarce. Beta-arrestins are proteins which inhibit G Protein Coupled Receptors and desensitize serotonergic and dopaminergic receptors. The study hypothesis is that Beta-arrestins 1 and 2 are predictive factors and biomarkers of response to antidepressants in major depressive disorder. In a controlled prospective open naturalistic monocentric 3-month study, 60 patients with a major depressive disorder requiring a treatment with venlafaxine will be included and assessed before treatment, 1 month and 3 months post-treatment. 20 controlled healthy subjects matched for age and gender will also be assessed. The Beta-arrestin pathway will be assessed using genetic polymorphisms, Peripheral Blood Mononuclear Cell measures and functional pathway. Antidepressant response will be assessed using depression scales, olfaction and memory as surrogate markers of neurogenesis.

DETAILED DESCRIPTION:
Rationale: Predictive factors and biomarkers of response to antidepressants in major depressive disorder are scarce. Beta-arrestins are proteins which inhibit G Protein Coupled Receptors and desensitize serotonergic and dopaminergic receptors.

Hypothesis: The study hypothesis is that Beta-arrestins 1 and 2 are predictive factors and biomarkers of response to antidepressants in major depressive disorder.

Method: In a controlled prospective open naturalistic monocentric 3-month study, 60 patients with a major depressive disorder requiring a treatment with venlafaxine will be included and assessed before treatment, 1 month and 3 months post-treatment. 20 controlled healthy subjects matched for age and gender will also be assessed.

Assessments:

The Beta-arrestin pathway will be assessed using genetic polymorphisms, Peripheral Blood Mononuclear Cell measures and functional pathway.

Antidepressant response will be assessed using depression scales, olfaction and memory as surrogate markers of neurogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Major Depressive Disorder
* current Major Depressive Episode
* Hamilton Depression Rating Scale score > 18
* requiring a new treatment with venlafaxine
* written informed consent

Exclusion Criteria:

* bipolar disorder
* psychotic disorder
* unstable somatic condition
* contraindication to cerebral RMI
* current treatment with mood stabilizers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-02-18 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in depressive symptoms on the Hamilton Depression Rating Scale-17 items | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle Corruble, MD, PhD, Principal Investigator — Inserm U669, APHP
Locations (1):
- CHU de Bicetre, Le Kremlin-Bicêtre, France

REFERENCES:
- [Background] Colle R, El Asmar K, Verstuyft C, Lledo PM, Lazarini F, Chappell K, Deflesselle E, Ait Tayeb AEK, Falissard B, Duron E, Rotenberg S, Costemale-Lacoste JF, David DJ, Gressier F, Gardier AM, Hummel T, Becquemont L, Corruble E. The olfactory deficits of depressed patients are restored after remission with venlafaxine treatment. Psychol Med. 2020 Oct 22:1-9. doi: 10.1017/S0033291720003918. Online ahead of print. PMID 33087184
- [Background] Baudouin E, Corruble E, Gori P, Bloch I, Becquemont L, Duron E, Colle R. White matter hyperintensities and their role in major depressive episodes: a cross-sectional study in adults under 65. Braz J Psychiatry. 2025;47:e20243921. doi: 10.47626/1516-4446-2024-3921. Epub 2024 Dec 28. PMID 39731725
- [Background] Mesdom P, Colle R, Becquemont L, Chappell K, David DJ, Mendez-David I, Corruble E, Verstuyft C. Tobacco use is associated with low peripheral beta-arrestin 1 levels in major depression: A preliminary report. Drug Alcohol Depend. 2022 Nov 1;240:109653. doi: 10.1016/j.drugalcdep.2022.109653. Epub 2022 Oct 2. PMID 36209675
- [Background] Etienne J, Boutigny A, David DJ, Deflesselle E, Gressier F, Becquemont L, Corruble E, Colle R. Habenular volume changes after venlafaxine treatment in patients with major depression. Psychiatry Clin Neurosci. 2024 Aug;78(8):468-472. doi: 10.1111/pcn.13684. Epub 2024 Jun 12. PMID 38867362
- [Background] Cussotto S, Colle R, Voican CS, Ciocan DM, Trainel N, Bottemanne H, Pelloux Y, David DJ, Cassard AM, Perlemuter G, Corruble E. The Gut Microbiota Is Altered in Antidepressant-Free Depressed Patients and Is Associated With Depression Severity. J Neurochem. 2025 Jul;169(7):e70173. doi: 10.1111/jnc.70173. PMID 40717539